CLINICAL TRIAL: NCT00851487
Title: A Randomized Multicentre Double Blind Trial of Amoxicillin Compared With Placebo for Treatment of WHO Defined Non-Severe Pneumonia in Children Aged 2-59 Months: NARIMA Study Group
Brief Title: Trial of Amoxicillin Compared With Placebo for Pneumonia in Children Aged 2-59 Months
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pakistan Institute of Medical Sciences (Other Government)
Collaborators: World Health Organization (Other)
Responsible Party: Dr. Tabish Hazir, ARI Research Cell, Children Hospital, PIMS, Islamabad
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NARIMA Study Group
Record Dates: First submitted 2009-02-25; First posted 2009-02-26 (Estimated); Last update posted 2009-02-26 (Estimated); Status verified 2009-02

CONDITIONS: Acute Respiratory Infections; Pneumonia
Keywords: ARI; LRTI
MeSH Terms: conditions — Pneumonia | interventions — Amoxicillin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Amoxicillin (Experimental): Oral amoxicillin in the dose of 15 mg/kg/dose 8 hourly was given as an active drug
  Interventions: Drug: Amoxicillin
- Placebo (Placebo Comparator): The placebo was similar in colour, consistency and volume as oral amoxicillin
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Amoxicillin — Oral Amoxicillin 15 mg/kg/dose 8 hourly
  Other Names: Amoxycillin
  Arms: Amoxicillin
Drug: Placebo — The placebo was similar in colour, consistency and volume as oral amoxicillin
  Arms: Placebo

SUMMARY:
Many children with "non-severe pneumonia" (cough and fast breathing) have neither clinical pneumonia as assessed by physicians nor pneumonia on chest radiographs. Inappropriate use of antibiotics for these cases is leading to resistant strains of bacteria in the community. Evidence shows that almost 50% of antibiotic prescription is unnecessary.As over half of antibiotic prescription for ARI are not necessary since most of these infections are viral and do not respond to antibiotic therapy which will be source of resistance in the community.

To address this issue the investigators conducted this randomized, double blind placebo controlled clinical trial of oral Amoxicillin versus placebo in children with non-severe pneumonia taking into account all the necessary safety precautions for their well being.

The study hypothesis was that the clinical outcome of children 2 to 59 months of age with cough and fast breathing (WHO defined non-severe pneumonia) with or without wheezing is equivalent, whether they are treated with amoxicillin or placebo.

DETAILED DESCRIPTION:
Pneumonia is one of the major cause of childhood morbidity and mortality in developing countries. Burden of acute respiratory infections (ARI) is high with an estimated 5-7 episodes in under 5 population every year resulting in 2 million deaths. However, most of these are due to severe bacterial pneumonia.

In order to reduce pneumonia related deaths in communities where qualified personnel and diagnostic facilities are often not available WHO developed management guidelines based on simple clinical signs followed by empirical treatment. All children with cough and fast breathing are classified into management categories: Children with fast breathing only are classified as having non-severe pneumonia requiring oral antibiotic at home, children who have lower chest indrawing and /or general danger signs (GDS) are classified as severe pneumonia, and very severe pneumonia respectively. Both these groups require referral to a hospital and injectible antibiotic therapy. These guidelines have shown to effectively reduce ARI related mortality by 34% (?) in communities where they have been successfully implemented.

However, there are certain concerns regarding these guidelines. It is felt that using the sign of fast breathing alone for prescribing antibiotic may not be the most judicious thing from a public health perspective as it may lead to the spread of antibiotic resistance. Fast breathing could be due to many other causes not related to pneumonia.

There are many factors affecting the respiratory rate I children. Children with fever will have elevated respiratory rates in any case. Although WHO guidelines recommend that respiratory rate must be counted when child is afebrile, calm and preferably sleeping. In real life such practice is not always possible.

Another issue is the children with cough and fast breathing who have wheezing. In many developing countries wheeze is commonly associated with fast and difficult breathing. Data from the developed countries shows that wheeze is more common in viral than bacterial infections. Likewise, data from the developing countries has shown that viruses, especially respiratory syncytial virus (RSV), are isolated more frequently than bacteria from children with episodes of acute lower respiratory tract infections. A randomized trial of infants with bronchiolitis and pneumonia found no difference in clinical outcome in children with antibiotics compared with placebo(ref?). Wheeze has long been unaddressed and is one of the major cause for overuse of antibiotics. Evidence shows that three cycles of inhaled bronchodilator was found to be associated with a significant decrease in respiratory rate leading to revised classification of "no pneumonia" in these children. It has convincingly shown that majority of these children continue to do well when sent home without an antibiotic.

Though fast breathing is an important indicator for clinical diagnosis of pneumonia it cannot distinguish viral from bacterial pathogens Controversy still exists concerning the relative importance of viral and bacterial pathogens so a reliable distinction between bacterial and viral infection has yet to be established and this issue has raised a lot of questions for the programme managers, senior researchers and technical experts, which still need to be answered.

Many children with "non-severe pneumonia" (cough and fast breathing) have neither clinical pneumonia as assessed by physicians nor pneumonia on chest radiographs. Inappropriate use of antibiotics for these cases is leading to resistant strains of bacteria in the community. Evidence shows that almost 50% of antibiotic prescription is unnecessary. As over half of antibiotic prescription for ARI are not necessary since most of these infections are viral and do not respond to antibiotic therapy which will be source of resistance in the community. When resistant bacteria become common, we may begin to see treatment failures in the children with severe pneumonia who really require an effective antibiotic. It is imperative to have the knowledge of likely cause and pattern of pneumonia which could be utilized to better understand the model of antibiotic resistance.

For the above stated reasons, there is a need to further elaborate the role of antibiotics in children with cough and fast breathing. To address this issue we conducted this randomized, double blind placebo controlled clinical trial of oral Amoxicillin versus placebo in children with non-severe pneumonia taking into account all the necessary safety precautions for their well being. The primary objective was to determine whether children aged 2 to 59 months with cough and fast breathing, with or without wheezing, but no evidence of WHO defined severe illness, have equivalent clinical failure at 72 hours of therapy when treated with Amoxicillin compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 2 to 59 months attending the outpatient's clinics of participating sites
* WHO defined non-severe pneumonia
* Accessibility for follow-up
* Written informed consent by a parent or legal guardian

Exclusion Criteria:

* WHO signs of severe pneumonia recognised by lower chest wall retraction. Children who present with wheezing will be evaluated for lower chest wall indrawing after treatments with nebulised salbutamol. WHO signs of very severe disease/pneumonia defined as any of the following:

  1. Cyanosis
  2. Inability to drink
  3. Convulsions
  4. Abnormally sleepy or difficult to wake
* Severe malnutrition recognised by weight for age less than third percentile by the NCHS (National Child Health Statistics) growth chart and/or oedema (see chart).
* All patients with a previous history of 3 or more episodes of wheeze or diagnosed to have asthma.
* Known or clinically recognisable congenital heart disease with cyanosis or, congestive heart failure or cardiomegaly.
* Known or clinically recognisable acute/chronic organ system disorders including jaundice, nephrotic syndrome, severe anaemia manifested as extreme pallor etc.
* Other infectious conditions requiring antibiotic therapy at the day of contact including meningitis, tuberculosis, dysentery, osteomyelitis, septic arthritis etc.
* Children who have taken the appropriate doses of WHO-recommended dose of anti microbial drug for 48 hours prior to presentation.
* A history of hospitalization in the past 2 weeks
* Measles or a history of measles within the last month: Measles recognized by presence of fever with rash, and conjunctivitis.
* Prior enrolment in the current trial.
* Known penicillin allergy, including a history of rash, urticaria, or anaphylactic symptoms.
* The children living outside the municipal limits of the city who cannot be followed up.

Ages: 2 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 900 (Actual)
Dates: Start 2006-01; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure was treatment failure within the first 72 hours of therapy | 3 days

SECONDARY OUTCOMES:
The secondary outcome measure was treatment failure on the third follow-up (day 5) plus non-improvement | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Tabish Hazir, FCPS-Peds, Principal Investigator — Overall Head of Research Cell; Dr. Yusra Ashraf, MBBS, Study Director — Research Administrator to ARI Research Cell
Locations (1):
- ARI Research Cell, Children Hospital, PIMS, Islamabad, Federal Capital, Pakistan